CLINICAL TRIAL: NCT04416061
Title: The Role of a Private Hospital in Hong Kong Amid COVID-19 Pandemic: A Descriptive Study of Patients With SARS-CoV-2 RT-PCR Performed
Brief Title: The Role of a Private Hospital in Hong Kong Amid COVID-19 Pandemic
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Hong Kong Sanatorium & Hospital (Industry)
Responsible Party: Principal Investigator, Dr. Jonpaul ST Zee, Specialist in Infectious Disease, Hong Kong Sanatorium & Hospital
Other Study IDs: RC-2020-08
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects underwent COVID-19 test: Subjects who underwent COVID-19 test in HKSH during the study period
  Interventions: Diagnostic Test: COVID 19 Diagnostic Test

INTERVENTIONS:
Diagnostic Test: COVID 19 Diagnostic Test — COVID 19 Diagnostic Test

SUMMARY:
Hong Kong public healthcare system is facing tremendous pressure under the COVID-19 pandemic. As the virus spread in Hong Kong, Hong Kong Sanatorium & Hospital (HKSH) is one of the first private hospitals which immediately provide reliable and rapid COVID-19 test -- Reverse Transcription Polymerase Chain Reaction (RT-PCR). Early provision of the RT-PCR screening test for COVID-19 not only facilitates identification of COVID-19 but also contains the spread of the virus in the community and frontline medical staff.

Since description of role of private hospital in Hong Kong amid COVID-19 pandemic is lacking, this study will describe COVID-19 screening algorithm and methodology. A retrospective analysis on clinical characteristics, laboratory findings as well as outcome of patients who underwent COVID-19 test in HKSH is also performed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who underwent COVID-19 test in HKSH during the study period

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who underwent COVID-19 test in HKSH during the study period
Sampling Method: Probability Sample
Enrollment: 2510 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of asymptomatic subjects | 1 Feb 2020 until the 14th consecutive day without any local infection in Hong Kong
  Proportion of asymptomatic subjects (%) who underwent COVID 19 test

SECONDARY OUTCOMES:
Proportion of subjects with recent contact history | 1 Feb 2020 until the 14th consecutive day without any local infection in Hong Kong
  Proportion of subjects (%) with recent contact history
Proportion of subjects with recent travel history | 1 Feb 2020 until the 14th consecutive day without any local infection in Hong Kong
  Proportion of subjects (%) with recent travel history

CONTACTS AND LOCATIONS:
Overall Officials: Jonpaul Sze Tsing Zee, MBChB, Principal Investigator — Hong Kong Sanatorium & Hospital
Locations (1):
- Hong Kong Sanatorium & Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No